CLINICAL TRIAL: NCT01503372
Title: Pazopanib With 5-Fluorouracil, Leucovorin and Oxaliplatin (FLO) as 1st-line Treatment in Advanced Gastric Cancer; a Randomized Phase-II-study of the Arbeitsgemeinschaft Internistische Onkologie
Brief Title: FLO +/- Pazopanib as First-line Treatment in Advanced Gastric Cancer
Acronym: PaFLO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, P. C. Thuss-Patience, consultant physician, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PaFLO; 2010-024379-15 (EudraCT Number)
Record Dates: First submitted 2011-12-22; First posted 2012-01-04 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Advanced Gastric Cancer
MeSH Terms: interventions — pazopanib; Fluorouracil; Oxaliplatin; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: FLO + Pazopanib (Experimental)
  Interventions: Drug: Pazopanib; Drug: 5-FU, Oxaliplatin, Leukovorin (FLO)
- Arm B: FLO (Active Comparator)
  Interventions: Drug: 5-FU, Oxaliplatin, Leukovorin (FLO)

INTERVENTIONS:
Drug: Pazopanib — Adding Pazopanib to a standard chemotherapy consisting of FLO. 800 mg (2x400mg or 4x200mg) Pazopanib per day should be taken orally without food at least one hour before or two hours after a meal. Pazopanib will be given d1-14 each cycle (2 weeks cycles) with 12 cycles of chemotherapy FLO (d 1, each cycle). After 12 cycles chemotherapy FLO will be discontinued and Pazopanib will be given alone until disease progression
  Arms: Arm A: FLO + Pazopanib
Drug: 5-FU, Oxaliplatin, Leukovorin (FLO) — Oxaliplatin 85 mg/m2 2h iv Leucovorin 200mg/m2 2h - iv FU 2600mg/m2 24h iv q2w for 12 cycles

SUMMARY:
The prognosis of advanced gastric cancer and adenocarcinoma of the gastro-esophageal (GE) junction is poor. Even with modern chemotherapy the median survival ranges around 8-10 months.

Inhibition of neoangiogenesis seems to be a very promising approach in gastric cancer.

Vascular endothelial growth factor (VEGF) acts as one of the most potent stimulating agents of angiogenesis, and several strategies targeting the VEGF signaling pathway have been developed, including anti-VEGF antibodies, soluble receptors binding directly to VEGF ligand, anti-VEGF receptor (VEGFR) antibodies and VEGFR tyrosine kinase inhibitors. The breakthrough in the clinical development of anti-angiogenic therapy against colorectal cancer came in 2003 with a large prospective, randomized clinical trial of bevacizumab, a monoclonal antibody directed against VEGF. Anti-angiogenic therapy has introduced a highly effective, completely new mode of action in this area and is the new standard of care in advanced colorectal cancer.

The concept of VEGF inhibition is also very promising in gastric cancer. Bevacizumab was investigated in combination with irinotecan and cisplatin in a phase-II trial, including 47 patients with gastric and GE-junction carcinoma. Bevacizumab could safely be given and could improve time to tumor progression by 75% compared to historical controls. Several phase-II trials confirm the tolerability and promising efficacy of bevacizumab in gastric cancer (Bevacizumab + Docetaxel/Oxaliplatin; FOLFOX + Bevacizumab; Docetaxel/Cisplatin/Irinotecan + Bevacizumab). These results were so promising that randomized phase-III trials in the 1st-line and perioperative setting are under way (AVAGAST-trial: Cisplatin /Capecitabine +/- bevacizumab 1st line ; MAGIC-B-trial : ECX +/- bevacizumab perioperative).

Tyrosin kinase inhibitors which inhibit VEGF receptors and EGFR are also investigated in gastric cancer with promising efficacy. Pazopanib, an orally available tyrosine kinase inhibitor, selectively inhibits vascular endothelial growth factor receptors (VEGFR)-1, -2 and -3, c-kit and platelet derived growth factor receptor (PDGF-R), which results in inhibition of angiogenesis in tumors in which these receptors are upregulated. Pazopanib has the advantage of being an orally available anti-angiogenesis component.

Pazopanib shows promising activity in phase-II trials in renal cell cancer, breast cancer, soft tissue sarcoma and non small cell lung cancer. A phase-III trial of pazopanib in renal cell cancer (NCT00334282) is completed and resulted in the approval of Pazopanib for this disease. A phase-III trial in soft tissue sarcoma (NCT00753688) is currently performed.

In phase-I trials, pazopanib was investigated in combination with FOLFOX and Capecitabine/Oxaliplatin. FOLFOX could be administered in full dose with 800 mg pazopanib. In Cape/Ox, capecitabine had to be reduced to 850mg/m² bd.

5-FU- and oxaliplatin-based regimens are one of the established treatment standards for 1st-line therapy in metastatic gastric cancer. The efficacy of 5-FU, leukovorin and oxaliplatin (FLO) compared to 5-FU, cisplatin could be confirmed in a randomized phase-III trial of the Arbeitsgemeinschaft Internistische Onkologie (AIO). FLO has a favorable toxicity profile. In Germany, FLO is a widely used combination for advanced gastric cancer and is a recommended regimen in the new German S3-guidelines 2011.

The investigators therefore want to examine FLO + pazopanib.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must provide written informed consent prior to performance of study-specific procedures or assessments, and must be willing to comply with treatment and follow up.
* Age ≥ 18 years.
* Histologically confirmed adenocarcinoma of the stomach or the gastroesophageal junction with either metastatic or locally advanced disease, incurable by operation.
* Eastern Cooperative Oncology Group (ECOG) performance status of < or = 2
* At least one unidimensional, measurable tumor parameter (according to RECIST 1.1)
* No preceding cytotoxic therapy (neoadjuvant or adjuvant treatment allowed if finished > 6 months before inclusion)
* Adequate organ system function.
* Men and women must perform an adequate contraception.
* Female subjects who are lactating should discontinue nursing prior to the first dose of study drug and should refrain from nursing throughout the treatment period and for 14 days following the last dose of study drug.

Exclusion Criteria:

* Prior malignancy, except for curatively treated basal cell carcinoma of the skin and in situ carcinoma of the cervix.
* Overexpression of HER-2, defined as IHC 3+ or IHC 2+ and FISH positive.
* Known hypersensitivity against 5-FU, leukovorin, oxaliplatin or other platinum compounds or pazopanib.
* History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis.
* Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding or the absorption of investigational product
* Presence of uncontrolled infection.
* Corrected QT interval (QTc) > 480 ms using Bazett's formula.
* History of any one or more of the following cardiovascular conditions within the past 6 months: cardiac angioplasty or stenting, myocardial infarction, unstable angina, coronary artery bypass graft surgery, symptomatic peripheral vascular disease, NYHA III or IV congestive heart failure.
* Poorly controlled hypertension.
* History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months.
* Prior major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer.
* Evidence of active bleeding or bleeding diathesis.
* Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels.
* Hemoptysis in excess of 2.5 ml within 8 weeks of first dose of study drug.
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures.
* Unable or unwilling to discontinue use of prohibited medications for at least 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of study drug and for the duration of the study.
* Treatment with any of the following anti-cancer therapies: radiation therapy, surgery or tumor embolization within 14 days prior to the first dose of pazopanib OR chemotherapy, immunotherapy, biologic therapy, investigational therapy or hormonal therapy within 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of pazopanib. A neoadjuvant or adjuvant chemotherapy must be finished at least 6 month before study entry.
* Any ongoing toxicity from prior anti-cancer therapy that is >Grade 1 and/or that is progressing in severity, except alopecia.
* Grade 3 or 4 diarrhea.
* Peripheral polyneuropathy > NCI Grade.
* Pregnant or lactating women.
* Men or women who are planning a pregnancy within the next six months.
* Participation in another clinical trial with investigational agents within the last 30 days prior to study start.
* The patient is a colleague or employed by the study investigator or by an involved institution including the sponsor of the study.
* Patient is detained in a psychiatric unit or imprisoned.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-11; Primary Completion 2017-12-14 (Actual); Study Completion 2017-12-14 (Actual)

PRIMARY OUTCOMES:
progression-free survival rate at 6 months | 6 months after study entry

SECONDARY OUTCOMES:
progression-free survival rate at 9 and 12 months | 9 and 12 months after study entry
median progression-free survival | 48 months
response rate | 48 months
duration of response | 48 months
toxicity | 48 months
  number of patients with Adverse Events according to CTC-criteria
tolerability | 48 months
  number of patients having adverse events and require interruptions and dose reductions of chemotherapy
overall survival | 48 months
time to treatment failure | 48 months
evaluation of the predictive and prognostic relevance of biomarkers | 48 months
  collection of plasma samples at designated time points during treatment and measuring of angiogenic factors correlating with response rate and outcome

CONTACTS AND LOCATIONS:
Overall Officials: Peter Thuss-Patience, MD, Study Chair — Charite University medicine
Locations (1):
- Charite University medicine, Berlin, Germany

REFERENCES:
- [Background] Shah MA, Ramanathan RK, Ilson DH, Levnor A, D'Adamo D, O'Reilly E, Tse A, Trocola R, Schwartz L, Capanu M, Schwartz GK, Kelsen DP. Multicenter phase II study of irinotecan, cisplatin, and bevacizumab in patients with metastatic gastric or gastroesophageal junction adenocarcinoma. J Clin Oncol. 2006 Nov 20;24(33):5201-6. doi: 10.1200/JCO.2006.08.0887. PMID 17114652
- [Background] El-Rayes BF, Patel B, Zalupski M, et al. A phase II study of bevacizumab, docetaxel, and oxaliplatin in gastric and GEJ cancer. ASCO Meeting Abstracts. 2009;27(15S):4563.
- [Background] Li J, Kortmansky JS, Saif M, et al. Phase II study of mFOLFOX6 with bevacizumab (Bev) in metastatic gastric and esophageal (GE) adenocarcinoma. ASCO Meeting Abstracts. 2010;28(15_suppl):TPS203.
- [Background] Enzinger PC, Ryan DP, Regan EM, et al. Phase II trial of docetaxel, cisplatin, irinotecan, and bevacizumab in metastatic esophagogastric cancer. ASCO Meeting Abstracts. 2008;26(15_suppl):4552.
- [Background] Sun W, Powell M, O'Dwyer PJ, Catalano P, Ansari RH, Benson AB 3rd. Phase II study of sorafenib in combination with docetaxel and cisplatin in the treatment of metastatic or advanced gastric and gastroesophageal junction adenocarcinoma: ECOG 5203. J Clin Oncol. 2010 Jun 20;28(18):2947-51. doi: 10.1200/JCO.2009.27.7988. Epub 2010 May 10. PMID 20458043
- [Background] Moehler MH, Hartmann JT, Lordick F, et al. An open-label, multicenter phase II trial of sunitinib for patients with chemorefractory metastatic gastric cancer. ASCO Meeting Abstracts. 2010;28(15_suppl):e14503.
- [Background] Hutson TE, Davis ID, Machiels JP, et al. Pazopanib (GW786034) is active in metastatic renal cell carcinoma (RCC): Interim results of a phase II randomized discontinuation trial (RDT). ASCO Meeting Abstracts. 2007;25(18_suppl):5031.
- [Background] Slamon D, Gomez HL, Kabbinavar FF, et al. Randomized study of pazopanib + lapatinib vs. lapatinib alone in patients with HER2-positive advanced or metastatic breast cancer. ASCO Meeting Abstracts. 2008;26(15_suppl):1016.
- [Background] Sleijfer S, Papai Z, Le Cesne A, et al. Phase II study of pazopanib (GW786034) in patients (pts) with relapsed or refractory soft tissue sarcoma (STS): EORTC 62043. ASCO Meeting Abstracts. 2007;25(18_suppl):10031.
- [Background] Altorki N, Guarino M, Lee P, et al. Preoperative treatment with pazopanib (GW786034), a multikinase angiogenesis inhibitor in early-stage non-small cell lung cancer (NSCLC): A proof-of-concept phase II study. ASCO Meeting Abstracts. 2008;26(15_suppl):7557.
- [Background] Brady J, Middleton M, Midgley RS, et al. A phase I study of pazopanib in combination with FOLFOX 6 or capeOx in subjects with colorectal cancer. ASCO Meeting Abstracts. 2009;27(15S):4133.
- [Background] Cunningham D, Starling N, Rao S, Iveson T, Nicolson M, Coxon F, Middleton G, Daniel F, Oates J, Norman AR; Upper Gastrointestinal Clinical Studies Group of the National Cancer Research Institute of the United Kingdom. Capecitabine and oxaliplatin for advanced esophagogastric cancer. N Engl J Med. 2008 Jan 3;358(1):36-46. doi: 10.1056/NEJMoa073149. PMID 18172173
- [Background] Al-Batran SE, Hartmann JT, Probst S, Schmalenberg H, Hollerbach S, Hofheinz R, Rethwisch V, Seipelt G, Homann N, Wilhelm G, Schuch G, Stoehlmacher J, Derigs HG, Hegewisch-Becker S, Grossmann J, Pauligk C, Atmaca A, Bokemeyer C, Knuth A, Jager E; Arbeitsgemeinschaft Internistische Onkologie. Phase III trial in metastatic gastroesophageal adenocarcinoma with fluorouracil, leucovorin plus either oxaliplatin or cisplatin: a study of the Arbeitsgemeinschaft Internistische Onkologie. J Clin Oncol. 2008 Mar 20;26(9):1435-42. doi: 10.1200/JCO.2007.13.9378. PMID 18349393
- [Background] Moehler M, Al-Batran SE, Andus T, Anthuber M, Arends J, Arnold D, Aust D, Baier P, Baretton G, Bernhardt J, Boeing H, Bohle E, Bokemeyer C, Bornschein J, Budach W, Burmester E, Caca K, Diemer WA, Dietrich CF, Ebert M, Eickhoff A, Ell C, Fahlke J, Feussner H, Fietkau R, Fischbach W, Fleig W, Flentje M, Gabbert HE, Galle PR, Geissler M, Gockel I, Graeven U, Grenacher L, Gross S, Hartmann JT, Heike M, Heinemann V, Herbst B, Herrmann T, Hocht S, Hofheinz RD, Hofler H, Hohler T, Holscher AH, Horneber M, Hubner J, Izbicki JR, Jakobs R, Jenssen C, Kanzler S, Keller M, Kiesslich R, Klautke G, Korber J, Krause BJ, Kuhn C, Kullmann F, Lang H, Link H, Lordick F, Ludwig K, Lutz M, Mahlberg R, Malfertheiner P, Merkel S, Messmann H, Meyer HJ, Monig S, Piso P, Pistorius S, Porschen R, Rabenstein T, Reichardt P, Ridwelski K, Rocken C, Roetzer I, Rohr P, Schepp W, Schlag PM, Schmid RM, Schmidberger H, Schmiegel WH, Schmoll HJ, Schuch G, Schuhmacher C, Schutte K, Schwenk W, Selgrad M, Sendler A, Seraphin J, Seufferlein T, Stahl M, Stein H, Stoll C, Stuschke M, Tannapfel A, Tholen R, Thuss-Patience P, Treml K, Vanhoefer U, Vieth M, Vogelsang H, Wagner D, Wedding U, Weimann A, Wilke H, Wittekind C; AWMF; AWMF. [German S3-guideline "Diagnosis and treatment of esophagogastric cancer"]. Z Gastroenterol. 2011 Apr;49(4):461-531. doi: 10.1055/s-0031-1273201. Epub 2011 Apr 7. No abstract available. German. PMID 21476183
- [Derived] Hogner A, Al-Batran SE, Siveke JT, Lorenz M, Bartels P, Breithaupt K, Malfertheiner P, Homann N, Stein A, Glaser D, Tamm I, Hinke A, Vogel A, Thuss-Patience P; PaFLO investigators. Pazopanib with 5-FU and oxaliplatin as first line therapy in advanced gastric cancer: A randomized phase-II study-The PaFLO trial. A study of the Arbeitsgemeinschaft Internistische Onkologie AIO-STO-0510. Int J Cancer. 2022 Mar 15;150(6):1007-1017. doi: 10.1002/ijc.33864. Epub 2021 Nov 15. PMID 34741530